CLINICAL TRIAL: NCT02746432
Title: Insulin Therapy Reduce Post-Operative Inflammatory Response After Curative Colorectal Cancer Resection: Randomization Controlled Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Mazen Hassanain, Assistant Professor & Counsultant HPB and transplant Surgeon, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: KSULDRCCRCMH001
Record Dates: First submitted 2016-04-06; First posted 2016-04-21 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Colon Cancer
Keywords: CRC-Insulin
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): Routine intra operative saline infusion to be administered.pre-operation and timed assessment lab set to be obtained.
- Intervention group.Hyper insulinemic euglycemic clamp (Experimental): After obtaining a baseline preoperative lab set blood glucose value, 2 U/kg bolus of insulin to be administered IV followed by an infusion of 2 U/ kg/min.fiver - Ten minutes after starting the insulin (Human regular insulin) ) infusion, and when the blood glucose is <6.1 mmol /L (110 mg /dL). an Infusion of dextrose 20% supplemented with pottasium phosphate (30 mmol/L ) to be administered. In the operating room, blood glucose levels were measured every 5-15 minutes, and the dextrose infusion rate was adjusted to maintain arterial glycemia between 3.5 and 6.1 mmol/L (63-110 mg/dL). timed intra operative lab assessment to be obtained.
  Interventions: Drug: Hyper insulinemic euglycemic clamp

INTERVENTIONS:
Drug: Hyper insulinemic euglycemic clamp — After obtaining a baseline preoperative lab set blood glucose value, 2 U/kg bolus of insulin (Human regular insulin) to be administered IV followed by an infusion of 2 U/ kg/min.fiver - Ten minutes after starting the insulin infusion, and when the blood glucose is <6.1 mmol /L (110 mg /dL). an Infusion of dextrose 20% supplemented with pottasium phosphate (30 mmol/L ) to be administered. In the operating room, blood glucose levels were measured every 5-15 minutes, and the dextrose infusion rate was adjusted to maintain arterial glycemia between 3.5 and 6.1 mmol/L (63-110 mg/dL). timed intra operative lab assessment to be obtained.
  Arms: Intervention group.Hyper insulinemic euglycemic clamp

SUMMARY:
Research Problem:

Surgical stress induces inflammation and postoperative immuno-suppression, which are risk.

factors for both post-operative complication and possible disease recurrence. Colorectal cancer is in the top 5 malignancies in the Kingdome and the highest incidence in males. Recurrent disease locally or distally occurs in 35% of patients and is the leading cause of death in these patients. Despite the new era of laparoscopic surgery, still surgical stress is present and equally traumatic to the conventional open colorectal resection, earlier studies showed no major differences in post-operative inflammatory and immunological reactions. The previous studies revealed the anti-inflammatory effects of the hyper-insulinimic euglycemic therapy. Benefits observed in both major liver resection and in cardiac surgery. The anti-inflammatory effect reduced the surgical stress and postoperative inflammation.

The hypothesis is "Can intraoperative hyper-insulinimic euglycemic infusion reduce post operative inflammation and immunomodulation in colon cancer patients undergoing a curative surgery?"

Research methodology Triple blinded randomized controlled study with estimated sample size of 144 patients of non-metastatic colorectal cancer patients operated at King Saud University Medical city with a confirmed diagnosis of colon adenocarcinoma. Patients Consented will undergo computer randomization to receive intraoperative hyper-insulinimic normoglycemic infusion (experimental) or standardized insulin sliding scale and saline (control). A common preoperative and postoperative pathway with standardized management and pain control in both groups.

Outcomes will be measured via a battery of laboratory test consist of routine labs, inflammatory markers and immunological markers to be repeated at fixed timed intervals. All patients will be followed by regularly for 5 years.

Research objectives

Primary outcomes to examine:

* The anti-inflammatory effects of intraoperative hyper-insulinimic euglycemic therapy in patients undergoing colorectal cancer surgery.
* The immunomodulatory effect of intraoperative hyper-insulinimic euglycemic infusion

Secondary outcomes:

* Thirty days post-operative morbidity.
* Overall survival rate.
* Disease-free survival rate.

DETAILED DESCRIPTION:
Aim & hypothesis:

The aim is to investigate the effect of the same protocol in colorectal surgery and to further delineate the effect on perioperative inflammation, immunosuppression and clinical outcome. This is an original approach, as this protocol was never used in bowel surgery.

The hypothesis predicts a reduced inflammation and resulting immunomodulation due to the anti-inflammatory effect of hyper-insulinmic euglycimic infusion, and improved postoperative morbidity and oncological outcome.

Study Design and Participants:

With the approval of the ethics board at King Saud University Medical city (KSUMC) a triple blinded randomized controlled study of operable resectable CRC patients of consented to be randomized to receive hyperinsulinimic normoglycemic protocol (experimental) or standardized insulin sliding scale (control).

Sample Size estimation:

72 patients per group( total of 144) was calculated to be sufficient to detect a reduction in disease recurrence from 35 to 20 percent, with α=0•05 and power of 0.8.

Randomization:

Computer generated randomization

Blinding:

Triple blinded study. Patient to be kept blinded to which group he/she will be assigned to. An independent anesthesia team will manage the infusion and will not be involved in the patient care or the study analysis. Research assistant will collect all the data and samples and will be blinded to the therapy. Patients' follow up by primary surgeons will also be blinded to the intervention. Analysis to be done in blinded groups A & B.

Intervention:

Intraoperative Intravenous insulin and glucose. The anasthesia will be asked to prepare an insulin bag containing 1000 units in 1 liter normal saline , another bag of dextrose 20 % with 30 mmol KPO4/ liter will be supplied from the pharmacy.

In the Experimental therapy group, after obtaining a baseline preoperative blood glucose value, 2 U/kg bolus of insulin to be administered IV followed by an infusion of 2 mU/ kg/min. Ten minutes after starting the insulin infusion, and when the blood glucose is <6.1 mmol /L (110 mg /dL), dextrose 20% supplemented with phosphate (30 mmol/L ) is administered. In the operating room, blood glucose levels were measured every 15 minutes, and the dextrose infusion rate will be adjusted to maintain arterial glycemia between 3.5 and 6.1 mmol/L (63-110 mg/dL), according to this protocol. If Blood Glucose mg/dl Action <63 Stop insulin infusion.Give Dextrose 20% 10 ml recheck level in 10 minutes 63.0 - 110 Maintain current infusion rate 111 - 143 144 - 180 Increase infusion by 2 unit/hour >180 Increase infusion by 3 unit/hour

The blood glucose will be measured hourly for 24 hours in the ICU, and the dextrose infusion rate was modified by the attending nurse according to this protocol (attached).

Regarding the safety of the patient on the hyperinsulinemia arms glucocheck every 5-10 minutes using an arterial line. Ongoing dextrose 20% + KPO4 supplementation when glucocheck drops less than 110 and will be titrated aimed to maintain a glucocheck 63-110. If at any point of time patient reached sever hypoglycemia defined as 32.3 (1.8) or below the insulin drip will be stopped and the patient will be considered a dropout of the study. Resuscitation with dextrose and KPO4 will continue to achieve eu-glycemia again. An international expert in the insulin clamp will be conducting the first patients to assure the local team experience for extra assurance.

Glucose Level mg/dl 20% Dextrose infusion + 30 meq Kcl <63 + 15 ml/h & 20ml bolus & Call MD 63-74 +10 ml/h & 10 ml bolus 75-81 + 5ml/h 82-98 Maintain the rate 99-110 - 5ml/h 111-116 -10ml/h >126 - 50% of the current rate & Call MD

In the standard therapy group, blood glucose measurements will be performed before the induction of anesthesia,every 30 minutes during surgery, and hourly in the ICU for 24 hours. If the blood glucose was >6.1 mmol /L (110 mg /dL), an insulin infusion of 1 U/ h was started. This was then titrated according to the sliding scale (Attached), aiming at a blood glucose between 3.5 and 6.1 mmol / L (63-110 mg/dL) during surgery and 3.5 and 7.9 mmol /L (63-143 mg /dL) after surgery A common preoperative and postoperative pathway with standardized management and pain control to be implemented in both groups. In diabetic patients, the administration of oral hypoglycemic drugs will be discontinued 24 hours before surgery. If patients received insulin, the daily dose will be held the evening before surgery, and subcutaneous insulin will be administered using a sliding scale. Arterial blood glucose concentrations measured using the glucocheck. Human insulin to be administered using the concentration 100 U of insulin in 100 mL normal saline.

Assessments:

Baseline preoperative investigations, 2 hours into surgery and a day 1 post operative, day 3, day 5, and 1 month postoperative assessment consisting of : Routine lab work

* CBC differential,
* Urea & electrolytes.
* Liver function test. Inflammatory assessment
* TNF-alpha,
* IL-8,
* IL-6
* IL-10
* IL-1β
* IL-18
* IFNγ
* MIP1α
* MMP-8
* TGF beta
* C-reactive protein The cytokines analysis will be done using suspension bead array immunoassay with a Luminex 200 X-map instrument (Luminex Corp, Austin, TX, USA). Analysis of the cytokines was carried out using a Milliplex human cytokine kit following manufacturer's specifications (MPXHCYTO-60k, Millipore Corp, Bilerica, MA, USA). All samples were analyzed in duplicate and the kit had a sensitivity of 0.4 pg/mL. Concentrations were calculated from the standard curve generated by the MasterPlex QT 4.0 analysis software (MiraiBio Inc, Alameda, CA, USA). Immunomodulation Quantity and activity of CD4, CD8, T-Cells T-cell profile
* Activation
* Proliferation
* Functionality (Intracellular cytokines profile). NK-Cells Profile
* Proliferation
* Activation *The degree of perioperative inflammation is a dynamic process that differs according to the time. The number of lab test is intended to build a curve describing the patient inflammatory response and the effect of insulin on it. The cytokines analysis will be done at the research lab, and only very few test will be sent to the hospital lab. The amount of blood taken will be limited to the tests, in the OR the bloods are taken from a dedicated line to prevent any discard.

The degree of perioperative inflammation is a dynamic process that differs according to the time . The number of lab test are intended to build a curve describing the patient inflammatory response and the effect of insulin on it.

Postoperative morbidity Postoperative events is defined and graded as per attached tables . non-infectious morbidity:

Morbidity Description Hyperglycemia >10 mmol/L Hypoglycemia <2 mmol/L PONV ( post operative nausea and vomiting) Persistent beyond day 2 postoperative Bleeding Requiring surgical intervention Or Hemoglobin drop >4 mg/dL Cardiac event Symptomatic arrhythmia Blood troponin >0.5, with ECG changes Pleural effusion Tapping required for patient relief Abdominal Ascites: dyspnea or leaking through abdominal wall Acute renal failure Serum creatinine >2 x upper limit of normal Anastomotic Leak Radiological luminal contrast extravasation Clinical finding of localized or generalized peritonitis Feculent drainage from drains Need for urgent intervention

Infectious morbidity:

Morbidity Description Pneumonia Pneumonic or atelactic changes on chest radiographs with positive sputum culture Wound infection Erythema and indurations associated with positive bacterial culture Intra-abdominal Collection of pus in the abdomen with or without necrotic material Abscess associated with a positive bacterial culture Urinary tract infection Urinary symptoms with urine culture positive for bacterial growth >105 colony forming units/ml Central line sepsis Positive culture of the catheter tip >15 colony forming units in the presence of febrile episode.

Leakage Grading according to International study group of rectal cancer (ISREC)

Grade Type of leak A Anastomotic leakage requiring no active therapeutic intervention. B Anastomotic leakage requiring active therapeutic intervention but manageable without laparotomy.

C Anastomotic leakage requiring Laparotomy.

Overall Morbidity grading Full Scale Grades Definition Grade I: Any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic and radiological interventions.

Allowed therapeutic regimens are: drugs as antiemetics, antipyretics, analgetics, diuretics and electrolytes and physiotherapy. This grade also includes wound infections opened at the bedside.

Grade II: Requiring pharmacological treatment with drugs other than such allowed for grade I complications.

Blood transfusions and total parenteral nutrition are also included. Grade III: Requiring surgical, endoscopic or radiological intervention Grade III-a: intervention not under general anesthesia Grade III-b: intervention under general anesthesia Grade IV: Life-threatening complication (including CNS complications)‡ requiring IC/ICU-management Grade IV-a: single organ dysfunction (including dialysis) Grade IV-b: multi organ dysfunction Grade V: Death of a patient Suffix 'd': If the patients suffers from a complication at the time of discharge, the suffix "d" (for 'disability') is added to the respective grade of complication. This label indicates the need for a follow-up to fully evaluate the complication.

Survival outcomes:

As per the guidelines all our patients will undergo a routine colonoscopy at 1 year and then after depending on the results, also a CT scan at 1 year, and 3 years and 5 years.

Data privacy and management:

In cardiac surgery it was mainly directed towards postoperative complication only and graft survival. In liver resection the main outcome was postoperative liver dysfunction and the micro mechanism were related to glycogen storage that might have been the cause for earlier and faster hepatic recovery. In our study, it's the first time to correlate it with anastomotic leak mainly and oncological outcomes. The use of this therapy has not made it to the clinical side because more studies are needed to confirm its efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Documented CRC by histopathology

Exclusion Criteria:

* Patient not consenting to the study or refused.
* Metastatic disease at the time of diagnosis.
* Contraindications to insulin
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
The anti-inflammatory effects of intraoperative hyper-insulinimic euglycemic therapy in patients undergoing colorectal cancer surgery. | 1 month
  effect on Inflamatory profile namely levels of Tnf- Alpha , IL-8 , IL-6 , IL-10 , IL-1B,IL-18 , IFNγ, MIp1-Alpha , MMP-8 , TGF Beta , CRP

SECONDARY OUTCOMES:
The immunomodulatory effect of intraoperative hyper-insulinimic euglycemic infusion. | 1 month
  Change of CD4 , CD8 & T-cell , Quantity and activity

OTHER OUTCOMES:
Thirty days post-operative morbidity | 30 days
Overall survival rate | 5 years
Disease-free survival rate | 5 years
Thirty days post-operative mortality | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- King Saud University Medical City, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Oberhofer D, Rumenjak V, Lazic J, Vucic N. [Inflammatory indicators in patients after surgery of the large intestine]. Acta Med Croatica. 2006 Dec;60(5):429-33. Croatian. PMID 17217098
- [Background] Galizia G, Gemei M, Orditura M, Romano C, Zamboli A, Castellano P, Mabilia A, Auricchio A, De Vita F, Del Vecchio L, Lieto E. Postoperative detection of circulating tumor cells predicts tumor recurrence in colorectal cancer patients. J Gastrointest Surg. 2013 Oct;17(10):1809-18. doi: 10.1007/s11605-013-2258-6. Epub 2013 Jun 28. PMID 23813048
- [Background] Rahbari NN, Aigner M, Thorlund K, Mollberg N, Motschall E, Jensen K, Diener MK, Buchler MW, Koch M, Weitz J. Meta-analysis shows that detection of circulating tumor cells indicates poor prognosis in patients with colorectal cancer. Gastroenterology. 2010 May;138(5):1714-26. doi: 10.1053/j.gastro.2010.01.008. Epub 2010 Jan 25. PMID 20100481
- [Background] Law WL, Choi HK, Lee YM, Ho JW. The impact of postoperative complications on long-term outcomes following curative resection for colorectal cancer. Ann Surg Oncol. 2007 Sep;14(9):2559-66. doi: 10.1245/s10434-007-9434-4. Epub 2007 May 24. PMID 17522945
- [Background] Deng HP, Chai JK. The effects and mechanisms of insulin on systemic inflammatory response and immune cells in severe trauma, burn injury, and sepsis. Int Immunopharmacol. 2009 Oct;9(11):1251-9. doi: 10.1016/j.intimp.2009.07.009. Epub 2009 Jul 30. PMID 19647101
- [Background] Albacker T, Carvalho G, Schricker T, Lachapelle K. High-dose insulin therapy attenuates systemic inflammatory response in coronary artery bypass grafting patients. Ann Thorac Surg. 2008 Jul;86(1):20-7. doi: 10.1016/j.athoracsur.2008.03.046. PMID 18573392
- [Background] Sato H, Carvalho G, Sato T, Bracco D, Codere-Maruyama T, Lattermann R, Hatzakorzian R, Matsukawa T, Schricker T. Perioperative tight glucose control with hyperinsulinemic-normoglycemic clamp technique in cardiac surgery. Nutrition. 2010 Nov-Dec;26(11-12):1122-9. doi: 10.1016/j.nut.2009.10.005. Epub 2010 Jan 25. PMID 20097532
- [Background] Wu FP, Sietses C, von Blomberg BM, van Leeuwen PA, Meijer S, Cuesta MA. Systemic and peritoneal inflammatory response after laparoscopic or conventional colon resection in cancer patients: a prospective, randomized trial. Dis Colon Rectum. 2003 Feb;46(2):147-55. doi: 10.1007/s10350-004-6516-2. PMID 12576886
- [Background] Sato H, Lattermann R, Carvalho G, Sato T, Metrakos P, Hassanain M, Matsukawa T, Schricker T. Perioperative glucose and insulin administration while maintaining normoglycemia (GIN therapy) in patients undergoing major liver resection. Anesth Analg. 2010 Jun 1;110(6):1711-8. doi: 10.1213/ANE.0b013e3181d90087. Epub 2010 Apr 7. PMID 20375299
- [Background] Ogawa K, Hirai M, Katsube T, Murayama M, Hamaguchi K, Shimakawa T, Naritake Y, Hosokawa T, Kajiwara T. Suppression of cellular immunity by surgical stress. Surgery. 2000 Mar;127(3):329-36. doi: 10.1067/msy.2000.103498. PMID 10715990
- [Background] Khansari DN, Murgo AJ, Faith RE. Effects of stress on the immune system. Immunol Today. 1990 May;11(5):170-5. doi: 10.1016/0167-5699(90)90069-l. PMID 2186751
- [Background] Parkin DM, Bray F, Ferlay J, Pisani P. Global cancer statistics, 2002. CA Cancer J Clin. 2005 Mar-Apr;55(2):74-108. doi: 10.3322/canjclin.55.2.74. PMID 15761078
- [Background] Law WL, Poon JT, Fan JK, Lo OS. Survival following laparoscopic versus open resection for colorectal cancer. Int J Colorectal Dis. 2012 Aug;27(8):1077-85. doi: 10.1007/s00384-012-1424-8. Epub 2012 Feb 9. PMID 22318646
- [Background] Basse L, Jakobsen DH, Bardram L, Billesbolle P, Lund C, Mogensen T, Rosenberg J, Kehlet H. Functional recovery after open versus laparoscopic colonic resection: a randomized, blinded study. Ann Surg. 2005 Mar;241(3):416-23. doi: 10.1097/01.sla.0000154149.85506.36. PMID 15729063
- [Derived] Bellon F, Sola I, Gimenez-Perez G, Hernandez M, Metzendorf MI, Rubinat E, Mauricio D. Perioperative glycaemic control for people with diabetes undergoing surgery. Cochrane Database Syst Rev. 2023 Aug 1;8(8):CD007315. doi: 10.1002/14651858.CD007315.pub3. PMID 37526194